CLINICAL TRIAL: NCT01133847
Title: Reading ICARD: Interventions for Children With Attention and Reading Disorders
Brief Title: Interventions for Children With Attention and Reading Disorders
Acronym: ICARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Carolyn Denton, Professor - Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-09-0531; R01HD060617 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-31 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Attention Deficit Hyperactivity Disorder; Reading Disabilities
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia | interventions — Methylphenidate; Atomoxetine Hydrochloride; Guanfacine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intensive Reading Instruction (Experimental): Specialized phonologically-based reading instruction provided by well-trained tutors either individually (one-on-one) or to groups of two students for 45 minutes, four days per week, for 16 weeks. The instructional approach includes an individualized combination of published programs targeting word reading and decoding; reading fluency; and reading comprehension.
  Interventions: Behavioral: Intensive reading instruction
- ADHD Intervention (Experimental): Carefully-managed medication and behavioral parent training. Medication treatment begins with a four-week titration period, beginning with a trial of methylphenidate. If benefit is insufficient or side effects are intolerable, the physician may initiate a trial of mixed salt amphetamine, followed by either Atomoxetine or Guanfacine. When the optimum medication and dosage is determined the child returns for monthly medication maintenance visits until the end of the 16-week intervention period. Parent training consists of nine group sessions provided by a psychologist addressing ADHD and its treatment, principals of behavior modification, and evidence-supported practices for managing behavior.
  Interventions: Drug: Methylphenidate; Behavioral: Parent Training; Drug: Mixed Salt Amphetamine; Drug: Atomoxetine; Drug: Guanfacine
- Combined ADHD and Reading Instruction (Experimental): All interventions described in Reading Instruction and ADHD treatment arms:
  Phonologically-based reading instruction provided for 45 minutes, four days per week, for 16 weeks. Carefully-managed medication and behavioral parent training. Medication treatment begins with a trial of methylphenidate. If benefit is insufficient or side effects are intolerable, the physician may initiate a trial of mixed salt amphetamine, followed by either Atomoxetine or Guanfacine. When the optimum medication and dosage is determined the child returns for monthly medication maintenance visits until the end of the 16-week intervention period. Parent training consists of nine group sessions on parenting a child with ADHD.
  Interventions: Drug: Methylphenidate; Behavioral: Intensive reading instruction; Behavioral: Parent Training; Drug: Mixed Salt Amphetamine; Drug: Atomoxetine; Drug: Guanfacine

INTERVENTIONS:
Drug: Methylphenidate — Appropriate dosage to be individually determined; daily for 16 weeks
  Other Names: Concerta Extended Release; Ritalin
  Arms: ADHD Intervention; Combined ADHD and Reading Instruction
Behavioral: Intensive reading instruction — Individualized phonologically-based instruction delivered 4 days per week for 45 min. per day by a highly trained tutor.
  Arms: Combined ADHD and Reading Instruction; Intensive Reading Instruction
Behavioral: Parent Training — Nine sessions on parenting a child with ADHD
  Arms: ADHD Intervention; Combined ADHD and Reading Instruction
Drug: Mixed Salt Amphetamine — Appropriate dosage to be individually determined; daily for 16 weeks; prescribed only if child does not show a beneficial treatment response to Concerta
  Other Names: Adderall Extended Release (XR)
  Arms: ADHD Intervention; Combined ADHD and Reading Instruction
Drug: Atomoxetine — Appropriate dosage to be individually determined; daily for 16 weeks
  Other Names: Strattera
  Arms: ADHD Intervention; Combined ADHD and Reading Instruction
Drug: Guanfacine — Appropriate dosage to be individually determined; daily for 16 weeks
  Other Names: Intuniv
  Arms: ADHD Intervention; Combined ADHD and Reading Instruction

SUMMARY:
The objective of this randomized clinical trial is to address unanswered questions about the relative effectiveness of treatments for children with both Attention Deficit Hyperactivity Disorder (ADHD) and significant reading difficulties (RD). The study evaluates attentional and word reading outcomes for students with both conditions when provided with either (a) ADHD treatment alone, (b) RD treatment alone, or (c) the combination of ADHD and RD treatment.

DETAILED DESCRIPTION:
The objective of this randomized clinical trial is to address unanswered questions about the relative effectiveness of treatments for children with both Attention Deficit Hyperactivity Disorder (ADHD) and significant reading difficulties (RD). The study evaluates attentional and word reading outcomes for students with both conditions when provided with either (a) disorder-specific ADHD treatment (carefully managed medication + parent training), (b) disorder-specific RD treatment (intensive, individualized reading instruction), or (c) the combination of ADHD and RD treatment. The study aims to address the relative benefits of providing either disorder-specific ADHD or RD treatment alone and providing the combined treatment. The investigators hypothesize that the combined treatment approach will result in better outcomes in terms of both word reading/decoding and a reduction in ADHD symptoms than either of the disorder-specific treatments alone. Treatment will last for 16 weeks, with assessment prior to and following treatment and some measures collected regularly throughout the intervention periods.

ELIGIBILITY:
Inclusion Criteria:

1. Meet criteria for ADHD, Combined Type or ADHD, Predominantly Inattentive Type based on the Diagnostic Interview Schedule for Children, 4.0 (DISC) parent interview, Teacher baseline Swanson Nolan and Pelham Rating Scale (SNAP) endorses additional non-overlapping Inattentive symptoms with the parent DISC, which when combined with the parent ratings result in endorsement of 6 or more symptoms required for diagnosis by the Diagnostic and Statistical Manual.
2. Have at least 4 symptoms of inattention rated "Often" or "Very Often" on the teacher version of the SNAP-IV.
3. Have a standard score of 90 or lower on either the Woodcock-Johnson III Tests of Achievement Letter-Word Identification or Word Attack Subtests, or on the Basic Reading Skills Cluster
4. Attend a participating school in Grades 2-5
5. Have at least one parent or guardian who understands English well enough to participate in the behavioral parent training intervention.
6. Have a Full Scale OR Non-Verbal Intelligence Quotient (IQ) estimate higher than 70 based on the IQ Composite and Non-Verbal IQ estimate of the Kaufman Brief Intelligence Test (KBIT-2).

Exclusion Criteria:

1. Any documented or suspected bipolar disorder, severe psychosis, or other severe emotional disturbance, developmental disability, or autism.
2. Receipt of primary school reading instruction in a language other than English.
3. A history or presence of cardiovascular problems that would contraindicate stimulant treatment.
4. Chronic vocal tics.
5. Children will be excluded if they are taking a concomitant medication that has the potential to significantly affect their ADHD symptoms, that would be contraindicated to take along with the study medication, or if they have not been on a stable dose of a psychotropic medication long enough to fully assess the clinical outcome or tolerability.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2010-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A Denton, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Texas Health Science Center, Houston, Texas

REFERENCES:
- [Derived] Dvorsky M, Tamm L, Denton CA, Epstein JN, Schatschneider C. Trajectories of Response to Treatments in Children with ADHD and Word Reading Difficulties. Res Child Adolesc Psychopathol. 2021 Aug;49(8):1015-1030. doi: 10.1007/s10802-021-00815-y. Epub 2021 Mar 26. PMID 33772416

RESULTS

PARTICIPANT FLOW:
Groups:
- ADHD Treatment: Carefully-managed medication and behavioral parent training. Children began with a trial of extended release methylphenidate; if there was no benefit or the side effects were intolerable, this was followed by a trial of mixed salt amphetamine. if side effects of stimulants were intolerable, atomoxetine or guanfacine could be prescribed. Parent training was nine sessions provided by a psychologist addressing ADHD and its treatment, principles of behavior modification, and evidence-supported practices for managing behavior.
- Intensive Reading Instruction: Specialized phonologically-based reading instruction provided by well-trained tutors either individually (one-on-one) or to groups of two students for 45 minutes, four days per week, for 16 school weeks. Instruction was explicit and systematic, with extended opportunities to practice and apply skills in connected text with feedback. Interventionists used an individualized combination of published and unpublished programs targeting word reading and decoding, reading fluency, and reading comprehension, depending on students' needs documented in ongoing assessment.
- Combined ADHD Treatment and Reading Instruction: All interventions described in Reading Instruction and ADHD treatment arms: Phonologically-based reading instruction provided for 45 minutes, four days per week, for 16 school weeks provided concurrently with carefully-managed medication (methylphenidate, mixed salt amphetamine, atomoxetine or guanfacine) and behavioral parent training.
Period: Active Treatment Phase (Weeks 1-16)
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Started | 78 | 74 | 70
Completed | 73 | 73 | 67
Not Completed | 5 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 1 | 3
Period: Follow-Up Phase
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Started | 73 | 73 | 67
Completed | 72 | 70 | 60
Not Completed | 1 | 3 | 7
Not completed — Lost to Follow-up | 1 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are for our final analysis sample, consisting of all children randomized to each condition except for 1 in the ADHD arm, 1 in the Reading arm, and 4 in the Combined arm, who were excluded because upon ex post-facto review of records, they did not meet either ADHD, RD, or IQ inclusion criteria and had been included in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction | Total
Number analyzed (Participants) | 77 | 73 | 66 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 77 | 73 | 66 | 216
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 35 | 84
  Male | 52 | 49 | 31 | 132
Region of Enrollment [Number; unit: participants]
  United States | 77 | 73 | 66 | 216

OUTCOME MEASURES:

1. Primary Outcome: Swanson, Nolan, and Pelham Checklist for DSM-IV (SNAP)- Parent Rating of Inattention
Description: Rating Scale of ADHD symptomology completed by parents and teachers. Raters evaluate how well each DSM-IV (Diagnostic and Statistical Manual) ADHD symptom describes a child on a four-point Likert scale (0=Not at all, 1=Just a little, 2=Quite a bit, 3=Very much). The measure shows adequate internal consistency (.94) and test-retest reliability (Bussing et al., 2008; Gau et al., 2008).
Time Frame: 16 weeks (end of Active Treatment phase), and follow-up
Population: Six excluded from analyses (1 from ADHD Treatment , 1 from Intensive Reading Instruction , 4 from Combined ) because upon ex post-facto review of records, they did not meet inclusion criteria and had been included in error. Other reductions in numbers analyzed on this variable were due to missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 71 | 72 | 60
Units on a scale
  16-Week Outcomes | 1.1 (0.1) | 1.7 (0.1) | 1.0 (0.1)
  Follow-up Outcomes | 1.3 (0.1) | 1.6 (0.1) | 1.0 (0.1)

2. Primary Outcome: Swanson, Nolan, and Pelham Checklist for DSM-IV (SNAP)- Parent Rating of Hyperactivity-impulsivity
Description: as for outcome 1
Time Frame: 16 weeks (end of Active Treatment phase), and follow-up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 71 | 72 | 60
units on a scale
  16-Week Outcomes | 0.8 (0.1) | 1.3 (0.1) | 0.6 (0.1)
  Follow-up Outcomes: number analyzed (Participants) | 66 | 66 | 52
  Follow-up Outcomes | 0.9 (0.1) | 1.4 (0.1) | 0.7 (0.1)

3. Primary Outcome: Swanson, Nolan, and Pelham Checklist for DSM-IV (SNAP)- Teacher Rating of Inattention
Description: Rating Scale of ADHD symptomology completed by parents and teachers. Raters evaluate how well each DSM-IV ADHD symptom describes a child on a four-point Likert scale (0=Not at all, 1=Just a little, 2=Quite a bit, 3=Very much). The measure shows adequate internal consistency (.94) and test-retest reliability (Bussing et al., 2008; Gau et al., 2008).
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 71 | 63
Units on a scale
  16-week Outcomes | 1.2 (0.1) | 1.7 (0.1) | 1.4 (0.1)
  Follow-Up: number analyzed (Participants) | 65 | 65 | 51
  Follow-Up | 1.5 (0.1) | 1.9 (0.1) | 1.5 (0.1)

4. Primary Outcome: Swanson, Nolan, and Pelham Checklist for DSM-IV (SNAP)- Teacher Rating of Hyperactivity-impulsivity
Description: as for outcome 3
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: Six excluded from analyses (1 from ADHD Treatment , 1 from Intensive Reading Instruction , 4 from Combined) because upon ex post-facto review of records, they did not meet inclusion criteria and had been included in error. Other reductions in numbers analyzed on this variable were due to missing data.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 71 | 63
Units on a scale
  16-Week Outcomes | 0.7 (0.1) | 1.1 (0.1) | 0.8 (0.1)
  Follow-up: number analyzed (Participants) | 65 | 65 | 51
  Follow-up | 0.8 (0.1) | 1.1 (0.1) | 0.8 (0.1)

5. Primary Outcome: Wechsler Individual Achievement Test-III (WIAT-III) Word Reading Subtest
Description: The WIAT-III is an individually-administered test of academic achievement. In the Word Reading subtest students read a list of increasingly difficult words. Scores reported here are standardized scores with a mean of 100 and standard deviation of 15.
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: Six excluded from analyses (1 from ADHD Treatment , 1 from Intensive Reading Instruction , 4 from Combined ) because upon ex post-facto review of records, they did not meet inclusion criteria and had been included in error. Other discrepancies in numbers are due to missing data.
Measure: Least Squares Mean (Standard Error); unit: standardized scores, M=100, SD = 15
Groups:
- Combined ADHD Treatment and Reading Instruction: All interventions described in Reading Instruction and ADHD treatment arms:
  All interventions described in Reading Instruction and ADHD treatment arms: Phonologically-based reading instruction provided for 45 minutes, four days per week, for 16 school weeks provided concurrently with carefully-managed medication (methylphenidate, mixed salt amphetamine, atomoxetine or guanfacine) and behavioral parent training.
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores, M=100, SD = 15
  16-Week Outcomes | 76.9 (0.7) | 79.0 (0.7) | 79.9 (0.7)
  Follow-Up: number analyzed (Participants) | 71 | 68 | 59
  Follow-Up | 77.1 (0.8) | 78.1 (0.8) | 78.8 (0.8)

6. Primary Outcome: Wechsler Individual Achievement Test-III (WIAT-III) Pseudoword Decoding Subtest
Description: The WIAT-III is an individually-administered test of academic achievement. In the Pseudoword Decoding subtest students read a list of increasingly difficult nonsense words as a test of their ability to use phonics to decode unknown words. Scores reported here are standardized scores with a mean of 100 and standard deviation of 15. Higher scores represent a better outcome.
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standardized scores
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores
  16-Week Outcomes | 78.3 (1.0) | 83.8 (1.0) | 83.0 (1.1)
  Follow-Up: number analyzed (Participants) | 71 | 68 | 59
  Follow-Up | 77.1 (1.0) | 82.6 (1.1) | 81.9 (1.2)

7. Secondary Outcome: Wechsler Individual Achievement Test-III (WIAT-III) Reading Comprehension Subtest
Description: The WIAT-III is an individually-administered test of academic achievement. This subtest involves reading sentences and longer passages and then answering a set of literal and inferential comprehension questions about the text. Scores reported here are standardized scores with a mean of 100 and standard deviation of 15. Higher scores represent a better outcome.
Time Frame: Week 16, End of Active Treatment Phase
Population: Six excluded from analyses (1 from ADHD Treatment , 1 from Intensive Reading Instruction , 4 from Combined ) because upon ex post-facto review of records, they did not meet inclusion criteria and had been included in error.
Measure: Least Squares Mean (Standard Error); unit: standardized scores
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores | 88.27 (0.9) | 84.70 (0.9) | 86.35 (1.0)

8. Secondary Outcome: Dynamic Indicators of Basic Early Literacy Skills Oral Reading Fluency Subtest (DIBELS ORF)
Description: DIBELS ORF measures oral reading fluency in connected text. Students are presented with a passage on their grade level to read orally, and the score is the number of words of the passage read correctly in a one-minute period. Students in this study read two passages at each test administration, and the mean score for the two passages was the dependent variable analyzed. A research synthesis of studies reporting psychometric properties for DIBELS ORF determined that reliability coefficients in these studies exceeded .80 and that the measure demonstrated moderate to high concurrent and predictive validity across studies (Goffreda & DiPerna, 2010).
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: words read correctly per minute
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
words read correctly per minute
  16-Week Outcomes | 53.67 (30.3) | 50.71 (31.94) | 53.83 (33.5)
  Follow-Up: number analyzed (Participants) | 70 | 68 | 59
  Follow-Up | 63.06 (31.97) | 57.40 (31.06) | 59.05 (31.97)

9. Secondary Outcome: Test of Word Reading Efficiency (TOWRE) - Sight Word Efficiency
Description: The TOWRE Sight Word Efficiency subtest measures fluency of reading words in lists. The raw score is the number of words or nonwords identified correctly in 45 seconds. Standard scores with a mean of 100 and standard deviaion of 15 are reported here. Higher scores represent a better outcome.
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standardized scores
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores
  16-Week Outcomes: number analyzed (Participants) | 72 | 72 | 59
  16-Week Outcomes | 80.8 (0.82) | 82.7 (0.82) | 83.5 (0.87)
  Follow-Up: number analyzed (Participants) | 70 | 68 | 59
  Follow-Up | 83.57 (0.82) | 85.04 (0.84) | 84.15 (0.90)

10. Secondary Outcome: Test of Word Reading Efficiency (TOWRE) - Phonemic Decoding Efficiency
Description: The TOWRE Phonemic Decoding Efficiency measures the student's fluent decoding of nonsense words that follow the spelling rules of the English language. The raw score is the number of nonwords identified correctly in 45 seconds. Standardized scores with a mean of 100 and standard deviaion of 15 are reported here. Higher scores represent a better outcome.
Time Frame: Week 16 (End of Active Treatment Phase) and Follow-Up
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standardized scores
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores
  16-Week Outcomes | 80.4 (0.79) | 83.4 (0.79) | 82.9 (0.84)
  Follow-Up: number analyzed (Participants) | 70 | 68 | 59
  Follow-Up | 81.49 (0.83) | 84.50 (0.86) | 84.32 (0.92)

11. Secondary Outcome: Test of Silent Reading Fluency and Comprehension (TOSREC)
Description: The TOSREC measures sentence-level comprehension and silent reading fluency. It is a sentence verification task; children are presented with a list of sentences and must tell whether they are true or false. Items are based on common knowledge (e.g., All apples are blue). The raw score is the number of items answered correctly in 3 minutes. Standardized with a mean of 100 and standard deviation of 15 are reported here. Higher scores represent a better outcome.
Time Frame: Week 16, End of Active Treatment Phase
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standardized scores
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Number analyzed (Participants) | 72 | 72 | 63
standardized scores | 17.40 (0.7) | 17.70 (0.7) | 18.57 (0.75)

ADVERSE EVENTS:
Time Frame: 6 years
Description: Children who received ADHD treatment (ADHD, Combined arms) were systematically assessed through regular clinic visits, phone calls, and rating scales of side effects and functioning completed by parents and teachers. Children receiving Reading Instruction were observed by their tutors about 4 days/week.
  Total at-risk (total monitored) = total in each arm who received some intervention. Those not receiving intervention were presumed not at-risk for treatment-related Adverse Events (AEs).
Arm/Group | ADHD Treatment | Intensive Reading Instruction | Combined ADHD Treatment and Reading Instruction
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/74 | 0/68
Other Adverse Events (participants affected / at risk) | 3/71 | 1/74 | 5/68
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADHD Treatment (N=71) | Intensive Reading Instruction (N=74) | Combined ADHD Treatment and Reading Instruction (N=68)
Aggressive behaviors (Social circumstances) | 3 (3) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
There was some non-adherence, particularly for the ADHD treatment. Our oversampling of low income, African American children, although valuable in an understudied population, may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No